CLINICAL TRIAL: NCT04949490
Title: A Phase II, Open-label, Rollover Trial to Evaluate the Safety and Immunogenicity of One or Two Boosting Doses of Comirnaty or One Dose of BNT162b2s01 in BNT162-01 Trial Subjects, or Two Boosting Doses of Comirnaty in BNT162-04 Trial Subjects
Brief Title: A Trial Investigating the Safety and Effects of One or Two Additional Doses of Comirnaty or One Dose of BNT162b2s01 in BNT162-01 or BNT162-04 Trial Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BNT162-14; 2021-002387-50 (EudraCT Number)
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: Infections, Respiratory; Virus Diseases; Infection Viral; Vaccine Adverse Reaction; RNA Virus Infections; Protection Against COVID-19 and Infections With SARS-CoV-2; Prevention of COVID-19 disease
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Virus Diseases; RNA Virus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A, BNT162b2s01 30 μg (1 dose) (Experimental): Trial participants from BNT162-01 (excluding transplant participants from Cohort 13) who received two injections of 30 μg BNT162b2 (Comirnaty) in the parent trial received one booster injection of BNT162b2s01 on Day 1. Day 1 (baseline in this trial) must have occurred ≥24 weeks after the last BNT162b2 (Comirnaty) injection in the parent BNT162-01 trial.
  Interventions: Biological: BNT162b2s01
- Group A, BNT162b2 30 μg (1 dose) (Experimental): Trial participants from BNT162-01 (excluding transplant participants from Cohort 13) who received two injections of 30 μg BNT162b2 (Comirnaty) in the parent trial received one booster injection of BNT162b2 (Comirnaty) on Day 1. Day 1 (baseline in this trial) must have occurred ≥24 weeks after the last BNT162b2 (Comirnaty) injection in the parent BNT162-01 trial.
  Interventions: Biological: BNT162b2
- Group B, BNT162b2 30 μg (2 doses) (Experimental): Trial participants in either the trial BNT162-01 (excluding transplant participants from Cohort 13) or BNT162-04 who did not receive the full two vaccinations of 30 μg BNT162b2 (Comirnaty) in the respective parent trial were offered two injections of 30 μg BNT162b2 (Comirnaty) as per the conditional marketing authorization on Day 1 and Day 21. Day 1 (baseline in this trial) must have occurred ≥12 weeks after receiving the last BNT162 candidate vaccine in the respective parent BNT162-01 or BNT162-04 trial.
  Interventions: Biological: BNT162b2
- Group B transplant subjects, BNT162b2 30 μg (2 doses) (Experimental): Transplant trial participants from Cohort 13 of the trial BNT162-01 received one injection of 30 μg BNT162b2 (Comirnaty) on Day 1 which was followed 3 to 7 months afterward by a second injection of BNT162b2 (Comirnaty). Day 1 (baseline in this trial) must have occurred ≥12 weeks after receiving the last BNT162 candidate vaccine in the parent BNT162-01 trial.
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2s01 — intramuscular (IM) injection
  Arms: Group A, BNT162b2s01 30 μg (1 dose)
Biological: BNT162b2 — IM injection
  Other Names: Comirnaty
  Arms: Group A, BNT162b2 30 μg (1 dose); Group B transplant subjects, BNT162b2 30 μg (2 doses); Group B, BNT162b2 30 μg (2 doses)

SUMMARY:
Trial to evaluate the safety and immunogenicity of one or two boosting doses of Comirnaty or one dose of BNT162b2s01 (Variant of concern [VOC] strain B.1.351) in BNT162-01 trial participants, or two boosting doses of Comirnaty in BNT162-04 trial participants.

Trial participants from BNT162-01 who received two injections of 30 μg Comirnaty were randomized 2:1 to one booster injection (BNT162b2s01: Comirnaty). Trial participants in either the trial BNT162-01 or BNT162-04 who did not receive the full two vaccinations of 30 μg Comirnaty were offered two injections of 30 μg Comirnaty as per the conditional marketing authorization. All potential rollover volunteers must enroll in this trial within less than 18 months of their last injection of a BNT162 candidate vaccine in the parent BNT162-01 or BNT162-04 trials.

DETAILED DESCRIPTION:
Group A trial participants were randomized 2:1 to BNT162b2s01:Comirnaty. Group B trial participants were allocated to trial treatment without active randomization and selected participants were asked to participate in the detailed immunogenicity assessment based on their parent trial cohort.

ELIGIBILITY:
Inclusion Criteria:

* Had given informed consent by signing the informed consent form (ICF) before initiation of any trial-specific procedures.
* Were willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions (including those requested by the German and federal Governments, e.g., to follow good practices to reduce chances of spreading COVID 19), and other requirements of the trial.
* Have received BNT162 vaccine candidates in the BNT162-01 or BNT162-04 trials.
* Remained overall healthy (i.e., has not medically deteriorated significantly since participation in the parent trial, is not anticipated to die in the next 26 weeks, and is able to provide blood as specified by the trial without anticipated, deleterious medical consequences) in the clinical judgment of the investigator based on medical history and physical examination. Screening clinical laboratory tests are to assess the participants' "new baseline" unless required for eligibility. Note: in particular, caution should be used with a subject who has a history of cardiovascular disease, e.g., myocarditis, pericarditis, myocardial infarction, congestive heart failure, cardiomyopathy, or clinically significant arrhythmia.
* Agreed not to enroll in another trial of an IMP, starting after Visit 0 and continuously until Visit 5 (Day 50).
* Less than 18 months have passed since their last IMP injection in their parent trial.
* If they received 30 μg Comirnaty twice in the BNT162-01 trial, Visit 1 in this trial is ≥24 weeks after their last IMP injection, unless the subject is a Cohort 13 transplant subject of the BNT162-01 trial.
* If they received any other BNT162 vaccine candidate than Comirnaty in the BNT162-01 or BNT162-04 trial or are a Cohort 13 transplant subject, Visit 1 in this trial is ≥12 weeks after their last IMP injection.
* Have not been diagnosed with SARS-CoV-2 infection in the 12 weeks prior to day 1 (baseline). Participants who screen-fail on this criterion may be rescreened.

Exclusion Criteria:

* Have received any SARS-CoV-2 vaccine outside of the BNT162-01 or BNT162-04 trials.
* Have had a known allergy, hypersensitivity, or intolerance to the planned IMP including any excipients of the IMP.
* Have had a current febrile illness (body temperature ≥38.0°C) or other acute illness within 48 hours prior to day 1/IMP injection in this trial. Participants who screen-fail on this criterion may be rescreened.
* Have received a live or live attenuated vaccine within 30 days prior to day 1/IMP injection, or any other vaccination within 14 days prior to day 1/IMP injection. Participants who screen-fail on this criterion may be rescreened.
* Have had an ongoing AE assessed as related to any BNT162-01 or BNT162-04 trial vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (4):
- Germany (4):
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - University Hospital Frankfurt, Infectiology, Frankfurt
  - University Hospital Heidelberg, Clinical Pharmacology, Heidelberg
  - CRS Clinical Research Services Mannheim GmbH, Mannheim

REFERENCES:
- [Derived] Quandt J, Muik A, Salisch N, Lui BG, Lutz S, Kruger K, Wallisch AK, Adams-Quack P, Bacher M, Finlayson A, Ozhelvaci O, Vogler I, Grikscheit K, Hoehl S, Goetsch U, Ciesek S, Tureci O, Sahin U. Omicron BA.1 breakthrough infection drives cross-variant neutralization and memory B cell formation against conserved epitopes. Sci Immunol. 2022 Sep 16;7(75):eabq2427. doi: 10.1126/sciimmunol.abq2427. Epub 2022 Sep 16. PMID 35653438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This rollover study (BNT162-14) has enrolled BNT162-01 (NCT04380701) or BNT162-04 (NCT04537949) study participants meeting all inclusion/exclusion criteria defined in the study protocol.
  The first participant was enrolled on 26 JUL 2021. The last visit of the last participant was on 16 SEP 2022.
Pre-assignment Details: All enrolled participants were allocated to treatment. Participants of the Group B immunology subset are also included in the respective Group B arms. Overall a total of 137 participants were enrolled into this study (including the Group B immunology subset participants).
Groups:
- Group A Comirnaty: Study participants from BNT162-01 (excluding transplant participants from Cohort 13) who received two injections of 30 μg BNT162b2 (Comirnaty) received one booster injection of BNT162b2 (Comirnaty) on Day 1.
  BNT162b2: intramuscular (IM) injection
- Group A BNT162b2s01: Study participants from BNT162-01 (excluding transplant participants from Cohort 13) who received two injections of 30 μg BNT162b2 (Comirnaty) received one booster injection of BNT162b2s01 on Day 1.
  BNT162b2s01: IM injection
- Group B Non-transplant Participants: Study participants in either the study BNT162-01 (excluding transplant participants from Cohort 13) or BNT162-04 who did not receive the full two vaccinations of 30 μg BNT162b2 (Comirnaty) were offered two injections of 30 μg BNT162b2 (Comirnaty) as per the conditional marketing authorization on Day 1 and Day 21.
  BNT162b2: IM injection
- Group B Transplant Participants; Group B Immunology Subset Transplant Participants: Transplant study participants from Cohort 13 of the study BNT162-01 received one injection of 30 μg BNT162b2 (Comirnaty) on Day 1 which will be followed 3 to 7 months afterward by a second injection of BNT162b2 (Comirnaty).
  BNT162b2: IM injection
- Group B Immunology Subset Non-transplant Participants: Study participants in either the study BNT162-01 (excluding transplant study participants from Cohort 13) or BNT162-04 who did not receive the full two vaccinations of 30 μg BNT162b2 (Comirnaty) were offered two injections of 30 μg BNT162b2 (Comirnaty) as per the conditional marketing authorization on Day 1 and Day 21.
  BNT162b2: IM injection
Period: Group A and Group B
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group B Non-transplant Participants | Group B Transplant Participants | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants
Started | 21 | 44 | 61 | 11 | 0 (Data of the Group B immunology subset participants is presented as separated period for full transparency.) | 0 (Data of the Group B immunology subset participants is presented as separated period for full transparency.)
Completed | 21 | 44 | 60 | 9 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Non-study SARS-COV-2 vaccination | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Subset Group B Immunogenicity Evaluation
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group B Non-transplant Participants | Group B Transplant Participants | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants
Started | 0 (Group A participants are not included in the Subset of Group B for Immunogenicity Evaluation.) | 0 (Group A participants are not included in the Subset of Group B for Immunogenicity Evaluation.) | 0 (Not all Group B participants are included in the subset of Group B for immunogenicity evaluation. Data of the participants included in the immunology subset is presented in separate columns on the right.) | 0 (Not all Group B participants are included in the subset of Group B for immunogenicity evaluation. Data of the participants included in the immunology subset is presented in separate columns on the right.) | 22 (Data of the Group B immunology subset participants is presented as separated period for full transparency.) | 11 (Data of the Group B immunology subset participants is presented as separated period for full transparency.)
Completed | 0 | 0 | 0 | 0 | 21 | 9
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Non-study SARS-COV-2 vaccination | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group B Non-transplant Participants | Group B Transplant Participants | Total
Number analyzed (Participants) | 21 | 44 | 61 | 11 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 28 | 50 | 11 | 106
  >=65 years | 4 | 16 | 11 | 0 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per the planned analyses, totals were only calculated for participants in Group A and Group B, respectively.
  years
    Group A: number analyzed (Participants) | 21 | 44 | 0 | 0 | 65
    Group A | 53.91 (15.13) | 55.81 (15.20) |  |  | 55.19 (15.09)
    Group B: number analyzed (Participants) | 0 | 0 | 61 | 11 | 72
    Group B |  |  | 49.17 (16.72) | 50.88 (11.92) | 49.43 (16.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 29 | 5 | 63
  Male | 12 | 24 | 32 | 6 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 44 | 61 | 11 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 21 | 42 | 61 | 11 | 135
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 21 | 44 | 61 | 11 | 137
Weight [Mean (Standard Deviation); unit: kg] — Population: Per the planned analyses, totals were only calculated for participants in Group A and Group B, respectively.
  kg
    Group A: number analyzed (Participants) | 21 | 44 | 0 | 0 | 65
    Group A | 76.76 (10.80) | 76.73 (13.45) |  |  | 76.74 (12.57)
    Group B: number analyzed (Participants) | 0 | 0 | 61 | 11 | 72
    Group B |  |  | 76.79 (13.86) | 74.14 (10.93) | 76.38 (13.42)

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Participants in Each Treatment Group With at Least One Serious Adverse Event (SAE) or Adverse Events of Special Interest (AESIs)
Description: For treatment-emergent SAEs and AESIs (TESAEs, TEAESIs), the data refers to the interval "Dose 1 up to 28 days after Dose 1". For other SAEs and AESIs, the data refers to the interval "Dose 1 up to 26 weeks after Dose 1".
  A TESAE/TEAESI is defined as any SAE/AESI with an onset after the first IMP dose or worsened after the first IMP dose (if the SAE/AESI was present before the first administration of IMP). SAEs/AESIs with an onset date more than 28 days after the last administration of IMP will be considered as TESAE/TEAESI only if assessed as related to IMP by the investigator.
  Participants of the Group B immunology subset are also included in the respective Group B arms and therefore counted in more than one arm/group. Overall a total of 137 participants were enrolled into this study (including the Group B immunology subset participants).
Time Frame: Up to 26 weeks after the first IMP injection
Population: Safety set, i.e., all participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Group A Total: All Group A study participants, i.e., study participants from BNT162-01 (excluding transplant participants from Cohort 13) who received two injections of 30 μg BNT162b2 (Comirnaty), received one booster injection of BNT162b2s01 or BNT162b2 on Day 1.
  BNT162b2s01 and BNT162b2: IM injection
- Group B Total: All Group B study participants, i.e., transplant study participants from Cohort 13 of the study BNT162-01 who received one injection of 30 μg BNT162b2 (Comirnaty) on Day 1 which was followed 3 to 7 months afterward by a second injection of 30 μg BNT162b2, and non-transplant study participants from either the study BNT162-01 (excluding transplant participants from Cohort 13) or BNT162-04 who did not receive the full two vaccinations of 30 μg BNT162b2 were offered two injections of 30 μg BNT162b2 as per the conditional marketing authorization on Day 1 and Day 21.
  BNT162b2: IM injection
- Group B Immunology Subset Total: All Group B immunology subset study participants, i.e., transplant study participants from Cohort 13 of the study BNT162-01 who received one injection of 30 μg BNT162b2 (Comirnaty) on Day 1 which was followed 3 to 7 months afterward by a second injection of 30 μg BNT162b2, and non-transplant study participants from either the study BNT162-01 (excluding transplant participants from Cohort 13) or BNT162-04 who did not receive the full two vaccinations of 30 μg BNT162b2 were offered two injections of 30 μg BNT162b2 as per the conditional marketing authorization on Day 1 and Day 21.
  BNT162b2: IM injection
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Non-transplant Participants | Group B Transplant Participants | Group B Total | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants | Group B Immunology Subset Total
Number analyzed (Participants) | 21 | 44 | 65 | 61 | 11 | 72 | 22 | 11 | 33
Participants
  Any SAE | 0 | 2 | 2 | 1 | 4 | 5 | 0 | 4 | 4
  Any related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TESAE | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Any related TESAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any related AESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: The Number and Percentage of Participants With Solicited Local Reactions at the Injection Site Recorded up to 7 Days After Each IMP Injection for Group A and for a Selected Subset (Immunology Subset) of Group B Participants.
Description: Local reactions (pain, tenderness, erythema/redness, induration/swelling) were graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"; the guidance uses the Grades 1 (mild), 2 (moderate), 3 (severe), and 4 (potentially life-threatening). The reporting of local reactions was based on the participant's assessments via daily solicited reports in the participant diaries.
  Participants of the Group B immunology subset are part of the Group B. The 'Total' arms include all participants from the respective Group A and Group B immunology subset arms presented.
Time Frame: Group A: From Day 1 to Day 8; For Group B (except transplant participants): From Day 1 to Day 8 for Dose 1, and from Day 22 to Day 29 for Dose 2. For Group B transplant participants: From Day 1 to Day 8 for Dose 1, and up to 7 days after Dose 2.
Population: Safety set, i.e., all participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants | Group B Immunology Subset Total
Number analyzed (Participants) | 21 | 44 | 65 | 22 | 11 | 33
Participants
  Dose 1 up to 7 days after Dose 1: Number of participants with any local reaction | 20 | 41 | 61 | 21 | 10 | 31
  Dose 1 up to 7 days after Dose 1: Number of participants with any grade >= 3 local reaction | 1 | 2 | 3 | 3 | 1 | 4
  Dose 2 up to 7 days after Dose 2: Number of participants with any local reaction: number analyzed (Participants) | 0 | 0 | 0 | 22 | 11 | 33
  Dose 2 up to 7 days after Dose 2: Number of participants with any local reaction |  |  |  | 20 | 5 | 25
  Dose 2 up to 7 days after Dose 2: Number of participants with any grade >= 3 local reaction: number analyzed (Participants) | 0 | 0 | 0 | 22 | 11 | 33
  Dose 2 up to 7 days after Dose 2: Number of participants with any grade >= 3 local reaction |  |  |  | 4 | 0 | 4

3. Primary Outcome: The Number and Percentage of Participants With Solicited Systemic Reactions Recorded up to 7 Days After Each IMP Injection for Group A and for a Selected Subset (Immunology Subset) of Group B Participants.
Description: Systemic reactions (nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills and fever) were graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"; the guidance uses the Grades 1 (mild), 2 (moderate), 3 (severe), and 4 (potentially life-threatening). The reporting of systemic reactions was based on the participant's assessments via daily solicited reports in the participant diaries.
  Participants of the Group B immunology subset are part of the Group B. The 'Total' arms include all participants from the respective Group A and Group B immunology subset arms presented.
Time Frame: as for outcome 2
Population: Safety set, i.e., all participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants | Group B Immunology Subset Total
Number analyzed (Participants) | 21 | 44 | 65 | 22 | 11 | 33
Participants
  Dose 1 up to 7 days after Dose 1: Number of participants with any systemic reaction | 18 | 33 | 51 | 20 | 8 | 28
  Dose 1 up to 7 days after Dose 1: Number of participants with any grade >= 3 systemic reaction | 4 | 9 | 13 | 2 | 0 | 2
  Dose 2 up to 7 days after Dose 2: Number of participants with any systemic reaction: number analyzed (Participants) | 0 | 0 | 0 | 22 | 6 | 28
  Dose 2 up to 7 days after Dose 2: Number of participants with any systemic reaction |  |  |  | 17 | 4 | 21
  Dose 2 up to 7 days after Dose 2: Number of participants with any grade >= 3 systemic reaction: number analyzed (Participants) | 0 | 0 | 0 | 22 | 6 | 28
  Dose 2 up to 7 days after Dose 2: Number of participants with any grade >= 3 systemic reaction |  |  |  | 7 | 0 | 7

4. Primary Outcome: The Number and Percentage of Participants With at Least One Unsolicited TEAE Occurring up to 28 Days After IMP Injection in Each Treatment Group for Group A and for a Selected Subset (Immunology Subset) of Group B Participants
Description: A TEAE is defined as any AE with an onset after the first IMP injection or worsened after the first IMP injection (if the AE was present before the first administration of IMP). AEs with an onset date more than 28 days after the last administration of IMP will be considered as treatment-emergent only if assessed as related to IMP by the investigator.
  Participants of the Group B immunology subset are part of the Group B. The 'Total' arms include all participants from the respective Group A and Group B immunology subset arms presented.
Time Frame: Group A: Up to 28 days after Dose 1. Group B: Up to 28 days after Dose 1 and up to 28 days after Dose 2.
Population: Safety set, i.e., all participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants | Group B Immunology Subset Total
Number analyzed (Participants) | 21 | 44 | 65 | 22 | 11 | 33
Participants
  Dose 1 up to 28 days after Dose 1: Number of participants with any TEAE | 8 | 14 | 22 | 5 | 6 | 11
  Dose 1 up to 28 days after Dose 1: Number of participants with any grade >=3 TEAE | 1 | 1 | 2 | 0 | 0 | 0
  Dose 2 up to 28 days after Dose 2; Number of participants with any TEAE: number analyzed (Participants) | 0 | 0 | 0 | 22 | 11 | 33
  Dose 2 up to 28 days after Dose 2; Number of participants with any TEAE |  |  |  | 5 | 2 | 7
  Dose 2 up to 28 days after Dose 2; Number of participants with any grade >=3 TEAE: number analyzed (Participants) | 0 | 0 | 0 | 22 | 11 | 33
  Dose 2 up to 28 days after Dose 2; Number of participants with any grade >=3 TEAE |  |  |  | 0 | 0 | 0

5. Secondary Outcome: Neutralizing Antibody Titers From Reference Strain and SARS-CoV-2 Variant B.1.351
Description: For Group A participants and Group B participants (except transplant subjects). Non-transplant participants of the Group B immunology subset are also part of the respective Group B arm and therefore occurring in more than one arm/group. The 'Total' arm for Group A include all participants from the Group A arms/groups.
Time Frame: Group A: At baseline (Day 1) and Day 8 and at Week 4 Day 29), Week 12 (Day 85), and Week 26 (Day 182). Group B: At baseline (Day 1) and Day 8 and at Week 3 (Day 22), Week 4 (Day 29), Week 7 (Day 50), Week 12 (Day 85), and Week 26 (Day 182).
Population: Immunogenicity set, i.e., all participants who received at least one dose of IMP and have at least one post-baseline immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Non-transplant Participants | Group B Immunology Subset Non-transplant Participants
Number analyzed (Participants) | 21 | 44 | 65 | 61 | 22
Titer
  Response neutralizing antibody titers reference strain - Baseline (Day 1) | 21.4 [13.2 to 34.5] | 21.3 [15.3 to 29.6] | 21.3 [16.4 to 27.7] | 15.6 [11.5 to 21.0] | 13.3 [8.3 to 21.3]
  Response neutralizing antibody titers variant B.1.351 - Baseline (Day1): number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response neutralizing antibody titers variant B.1.351 - Baseline (Day1) | NA [NA to NA] — Titers were below lower limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers were below lower limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers were below lower limit of detection. Confidence intervals were not computable. |  |
  Response neutralizing antibody titers reference strain - Day 8 | 640.0 [376.6 to 1087.7] | 349.0 [254.5 to 478.6] | 424.5 [322.5 to 558.8] | 729.3 [485.4 to 1095.8] | 1093.4 [719.8 to 1661.0]
  Response neutralizing antibody titers variant B.1.351 - Day 8: number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response neutralizing antibody titers variant B.1.351 - Day 8 | 285.1 [164.2 to 495.0] | 330.2 [232.3 to 469.5] | 314.9 [235.8 to 420.6] |  |
  Response neutralizing antibody titers reference strain - Week 3 (Day 22): number analyzed (Participants) | 0 | 0 | 0 | 61 | 22
  Response neutralizing antibody titers reference strain - Week 3 (Day 22) |  |  |  | 1085.6 [775.5 to 1519.5] | 1183.0 [738.2 to 1896.0]
  Response neutralizing antibody titers reference strain - Week 4 (Day 29) | 570.2 [309.3 to 1051.1] | 509.3 [372.4 to 696.6] | 528.2 [399.1 to 699.2] | 1789.7 [1367.3 to 2342.6] | 1868.1 [1278.7 to 2729.3]
  Response neutralizing antibody titers variant B.1.351 - Week 4 (Day 29): number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response neutralizing antibody titers variant B.1.351 - Week 4 (Day 29) | 271.3 [157.9 to 466.1] | 325.1 [233.2 to 453.3] | 306.6 [232.4 to 404.6] |  |
  Response neutralizing antibody titers reference strain - Week 7: number analyzed (Participants) | 0 | 0 | 0 | 61 | 22
  Response neutralizing antibody titers reference strain - Week 7 |  |  |  | 1386.0 [1054.5 to 1821.6] | 1429.2 [864.5 to 2362.8]
  Response neutralizing antibody titers reference strain - Week 12 (Day 85): number analyzed (Participants) | 21 | 33 | 54 | 60 | 21
  Response neutralizing antibody titers reference strain - Week 12 (Day 85) | 371.2 [202.5 to 680.5] | 282.1 [181.0 to 439.8] | 313.9 [221.5 to 444.9] | 1348.3 [992.8 to 1831.1] | 1301.3 [795.2 to 2129.5]
  Response neutralizing antibody titers variant B.1.351 - Week 12 (Day 85): number analyzed (Participants) | 21 | 33 | 54 | 0 | 0
  Response neutralizing antibody titers variant B.1.351 - Week 12 (Day 85) | 122.9 [65.3 to 231.4] | 259.4 [162.6 to 413.7] | 194.0 [133.0 to 282.9] |  |
  Response neutralizing antibody titers reference strain - Week 26 (Day 182): number analyzed (Participants) | 21 | 18 | 39 | 57 | 20
  Response neutralizing antibody titers reference strain - Week 26 (Day 182) | 336.2 [159.6 to 708.6] | 132.0 [64.6 to 269.7] | 218.4 [130.0 to 366.8] | 659.8 [469.5 to 927.1] | 710.1 [439.5 to 1147.3]
  Response neutralizing antibody titers variant B.1.351 - Week 26 (Day 182): number analyzed (Participants) | 21 | 18 | 39 | 0 | 0
  Response neutralizing antibody titers variant B.1.351 - Week 26 (Day 182) | 140.2 [60.4 to 325.2] | 129.5 [63.8 to 262.6] | 135.1 [79.3 to 230.3] |  |

6. Secondary Outcome: Antibody Titers (ELISA) to Recombinant S1 and RBD Protein Derived From Reference and SARS-CoV-2 Variant B.1.351
Description: For Group A participants and Group B participants (except transplant subjects). Non-transplant participants in the Group B immunology subset arm are also part of the respective Group B arm and therefore occurring in more than one arm/group. The 'Total' arm for Group A include all participants from the Group A arms/groups.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Non-transplant Participants | Group B Immunology Subset Non-transplant Participants
Number analyzed (Participants) | 21 | 44 | 65 | 61 | 22
Titer
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Baseline (Day1) | 2216.1 [1507.6 to 3257.7] | 2161.4 [1634.7 to 2857.8] | 2178.9 [1748.0 to 2716.1] | 2135.4 [1303.7 to 3497.5] | 2056.4 [1297.3 to 3259.6]
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Baseline (Day 1): number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Baseline (Day 1) | 566.5 [370.9 to 865.3] | 588.7 [438.4 to 790.6] | 581.5 [459.5 to 735.8] |  |
  Response antibody titers IgG S Protein reference strain (ELISA) - Baseline (Day 1) | 3209.0 [2045.6 to 5033.9] | 2594.7 [1977.5 to 3404.4] | 2779.1 [2210.9 to 3493.2] | 1634.4 [1025.5 to 2605.0] | 1636.2 [885.2 to 3024.5]
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Baseline (Day 1): number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Baseline (Day 1) | 7164.8 [4231.7 to 12130.9] | 9267.9 [6837.3 to 12562.5] | 8528.4 [6572.5 to 11066.5] |  |
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Day 8 | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | 48945.7 [35518.9 to 67447.9] | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | 48805.7 [29759.0 to 80043.1] | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Day 8: number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Day 8 | 22903.0 [11936.4 to 43945.2] | 21244.0 [15712.2 to 28723.3] | 21766.4 [16403.7 to 28882.2] |  |
  Response antibody titers IgG S Protein reference strain (ELISA) - Day 8 | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | 45270.4 [27269.8 to 75153.2] | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Day 8: number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Day 8 | 520744.5 [258322.6 to 1049752.6] | 480042.7 [319790.9 to 720599.2] | 492832.1 [348924.0 to 696092.7] |  |
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 3: number analyzed (Participants) | 0 | 0 | 0 | 61 | 22
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 3 |  |  |  | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 3: number analyzed (Participants) | 0 | 0 | 0 | 61 | 22
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 3 |  |  |  | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 4 | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Week 4: number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Week 4 | 18959.7 [11062.8 to 32493.5] | 21082.1 [16052.9 to 27686.8] | 20371.6 [15940.0 to 26035.3] |  |
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 4 | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Week 4: number analyzed (Participants) | 21 | 44 | 65 | 0 | 0
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Week 4 | 394493.5 [198914.7 to 782371.2] | 362296.9 [259569.0 to 505680.9] | 372400.7 [274455.6 to 505299.6] |  |
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 7: number analyzed (Participants) | 0 | 0 | 0 | 61 | 22
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 7 |  |  |  | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 7: number analyzed (Participants) | 0 | 0 | 0 | 61 | 22
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 7 |  |  |  | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 12: number analyzed (Participants) | 21 | 33 | 54 | 60 | 21
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 12 | 23883.9 [15193.4 to 37545.2] | 28535.3 [20676.5 to 39381.0] | 26627.5 [20616.5 to 34391.0] | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Week 12: number analyzed (Participants) | 21 | 33 | 54 | 0 | 0
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Week 12 | 11106.8 [6446.7 to 19135.5] | 14367.3 [9798.4 to 21066.5] | 12998.8 [9570.3 to 17655.4] |  |
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 12: number analyzed (Participants) | 21 | 33 | 54 | 60 | 21
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 12 | 50709.2 [33710.6 to 76279.3] | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Week 12: number analyzed (Participants) | 21 | 33 | 54 | 0 | 0
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Week 12 | 178167.5 [95710.4 to 331663.8] | 305041.0 [196223.1 to 474205.2] | 247480.6 [173229.4 to 353558.0] |  |
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 26: number analyzed (Participants) | 21 | 18 | 39 | 57 | 20
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 26 | 14309.8 [7900.1 to 25920.0] | 8670.5 [5238.9 to 14349.9] | 11355.5 [7717.3 to 16709.0] | 34032.7 [25327.8 to 45729.3] | 38865.2 [23611.8 to 63972.6]
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Week 26: number analyzed (Participants) | 21 | 18 | 39 | 0 | 0
  Response antibody titers IgG RBD Domain variant B.1.351 (ELISA) - Week 26 | 9829.9 [4948.4 to 19526.7] | 6967.7 [4124.5 to 11770.9] | 8386.3 [5479.1 to 12835.9] |  |
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 26: number analyzed (Participants) | 21 | 18 | 39 | 57 | 20
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 26 | 27732.0 [15894.6 to 48385.3] | 17049.8 [10185.6 to 28539.8] | 22155.2 [15250.2 to 32186.6] | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable. | NA [NA to NA] — Titers above upper limit of detection. Confidence intervals were not computable.
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Week 26: number analyzed (Participants) | 21 | 18 | 39 | 0 | 0
  Response antibody titers IgG S Protein variant B.1.351 (ELISA) - Week 26 | 142683.7 [67849.2 to 300057.1] | 91825.4 [50843.9 to 165838.9] | 116420.8 [72901.4 to 185919.5] |  |

7. Secondary Outcome: SARS-CoV-2 Functional Cross-neutralization (GMT Ratios) of Variant B.1.351 to Reference Strain
Description: For Group A only. The geometric mean titer (GMT) ratio is calculated as the GMT of reference divided by the GMT of variant B.1.351.
  The 'Total' arm for Group A include all participants from the two Group A arms/groups.
Time Frame: Up to 26 weeks after the first IMP injection (Dose 1)
Population: as for outcome 5
Measure: Number; unit: GMT ratio
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total
Number analyzed (Participants) | 21 | 44 | 65
GMT ratio
  Day 1 - Response neutralizing antibody titers - GMT ratio | 3.1 | 3.0 | 3.0
  Day 1 - Response antibody titers IgG RBD Domain - GMT ratio | 3.9 | 3.7 | 3.7
  Day 1 - Response antibody titers IgG S Protein - GMT ratio | 0.4 | 0.3 | 0.3
  Day 8 - Response neutralizing antibody titers - GMT ratio | 2.2 | 1.1 | 1.3
  Day 8 - Response antibody titers IgG RBD Domain - GMT ratio | 2.9 | 2.3 | 2.5
  Day 8 - Response antibody titers IgG S Protein - GMT ratio | 0.2 | 0.2 | 0.2
  Week 4 (Day 29) - Response neutralizing antibody titers - GMT ratio | 2.1 | 1.6 | 1.7
  Week 4 (Day 29) - Response antibody titers IgG RBD Domain - GMT ratio | 3.1 | 2.6 | 2.8
  Week 4 (Day 29) - Response antibody titers IgG S Protein - GMT ratio | 0.2 | 0.2 | 0.2
  Week 12 (Day 85) - Response neutralizing antibody titers - GMT ratio: number analyzed (Participants) | 21 | 33 | 54
  Week 12 (Day 85) - Response neutralizing antibody titers - GMT ratio | 3.0 | 1.1 | 1.6
  Week 12 (Day 85) - Response antibody titers IgG RBD Domain - GMT ratio: number analyzed (Participants) | 21 | 33 | 54
  Week 12 (Day 85) - Response antibody titers IgG RBD Domain - GMT ratio | 2.2 | 2.0 | 2.0
  Week 12 (Day 85) - Response antibody titers IgG S Protein - GMT ratio: number analyzed (Participants) | 21 | 33 | 54
  Week 12 (Day 85) - Response antibody titers IgG S Protein - GMT ratio | 0.3 | 0.2 | 0.2
  Week 26 (Day 182) - Response neutralizing antibody titers - GMT ratio: number analyzed (Participants) | 21 | 18 | 39
  Week 26 (Day 182) - Response neutralizing antibody titers - GMT ratio | 2.4 | 1.0 | 1.6
  Week 26 (Day 182) - Response antibody titers IgG RBD Domain - GMT ratio: number analyzed (Participants) | 21 | 18 | 39
  Week 26 (Day 182) - Response antibody titers IgG RBD Domain - GMT ratio | 1.5 | 1.2 | 1.4
  Week 26 (Day 182) - Response antibody titers IgG S Protein - GMT ratio: number analyzed (Participants) | 21 | 18 | 39
  Week 26 (Day 182) - Response antibody titers IgG S Protein - GMT ratio | 0.2 | 0.2 | 0.2

8. Secondary Outcome: Neutralizing Antibody Titers (Reference Strain) Derived From SARS-CoV-2
Description: For Group B transplant subjects, assessed at baseline (Day 1 of Dose 1) and then Day 8, Weeks 4, 12, and 26 post Dose 1, and at Dose 2 (Day 1) and the Day 8, Weeks 4, 12, and 26 post Dose 2.
  Because the 11 participants of the arm 'Group B Immunology Subset Transplant Participants' are the same 11 participants of the arm 'Group B Immunology Subset Transplant Participants', data is not presented for this arm to avoid duplication of data.
Time Frame: From baseline (Day 1 of Dose 1) up to 26 weeks after Dose 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group B Transplant Participants
Number analyzed (Participants) | 11
Titer
  Day 1 of Dose 1 | NA [NA to NA] — Titers were below lower limit of detection. Confidence intervals were not computable.
  Day 8 of Dose 1 | 48.3 [13.0 to 179.2]
  Week 4 (Day 29) of Dose 1 | 124.4 [25.4 to 609.6]
  Week 12 (Day 85) of Dose 1 | 80.0 [17.1 to 374.8]
  Week 26 (Day 182) of Dose 1: number analyzed (Participants) | 9
  Week 26 (Day 182) of Dose 1 | 108.9 [23.1 to 513.0]
  Day 1 pre Dose 2: number analyzed (Participants) | 6
  Day 1 pre Dose 2 | 47.6 [7.3 to 311.5]
  Day 8 post Dose 2: number analyzed (Participants) | 6
  Day 8 post Dose 2 | 142.5 [9.4 to 2160.6]
  Week 4 (Day 29) post Dose 2: number analyzed (Participants) | 6
  Week 4 (Day 29) post Dose 2 | 452.5 [61.7 to 3317.6]
  Week 12 (Day 85) post Dose 2: number analyzed (Participants) | 6
  Week 12 (Day 85) post Dose 2 | 142.5 [21.5 to 945.6]
  Week 26 (Day 182) post Dose 2: number analyzed (Participants) | 6
  Week 26 (Day 182) post Dose 2 | 127.0 [19.7 to 819.1]

9. Secondary Outcome: Antibody Titers (ELISA) (Reference Strain) to Recombinant S1 and RBD Protein Derived From SARS-CoV-2
Description: as for outcome 8
Time Frame: From baseline (Day 1 of Dose 1) up to 26 weeks after Dose 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group B Transplant Participants
Number analyzed (Participants) | 11
Titer
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Baseline (Day 1 of Dose 1) | 730.5 [157.1 to 3397.0]
  Response antibody titers IgG S Protein reference strain (ELISA) - Baseline (Day 1 of Dose 1) | 599.1 [117.1 to 3064.9]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Day 8 of Dose 1 | 4328.8 [512.9 to 36532.1]
  Response antibody titers IgG S Protein reference strain (ELISA) - Day 8 of Dose 1 | 5078.0 [528.0 to 48838.3]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 4 (Day 29) of Dose 1 | 6616.9 [987.7 to 44327.3]
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 4 (Day 29) of Dose 1 | 7937.6 [1179.2 to 53431.0]
  Response antibody titers IgG RBD Domain reference strain (ELISA)- Week 12 (Day 85) of Dose 1 | 5065.9 [791.0 to 32443.1]
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 12 (Day 85) of Dose 1 | 11988.6 [1607.4 to 89413.3]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 26 (Day 182) of Dose 1: number analyzed (Participants) | 9
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 26 (Day 182) of Dose 1 | 10602.6 [2076.7 to 54130.4]
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 26 (Day 182) of Dose 1: number analyzed (Participants) | 9
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 26 (Day 182) of Dose 1 | 19644.7 [5085.2 to 75890.1]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Day 1 pre Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Day 1 pre Dose 2 | 3633.0 [506.1 to 26078.1]
  Response antibody titers IgG S Protein reference strain (ELISA) - Day 1 pre Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG S Protein reference strain (ELISA) - Day 1 pre Dose 2 | 5822.9 [894.5 to 37904.8]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Day 8 post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Day 8 post Dose 2 | 12441.7 [1398.3 to 110702.9]
  Response antibody titers IgG S Protein reference strain (ELISA) - Day 8 post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG S Protein reference strain (ELISA) - Day 8 post Dose 2 | 22067.6 [2752.2 to 176945.0]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 4 (Day 29) post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 4 (Day 29) post Dose 2 | 13625.0 [2884.8 to 64350.9]
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 4 (Day 29) post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 4 (Day 29) post Dose 2 | 34242.9 [7476.0 to 156845.8]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 12 (Day 85) post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 12 (Day 85) post Dose 2 | 12265.4 [1706.1 to 88179.1]
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 12 (Day 85) post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 12 (Day 85) post Dose 2 | 24015.7 [3852.9 to 149692.4]
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 26 (Day 182) post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG RBD Domain reference strain (ELISA) - Week 26 (Day 182) post Dose 2 | 13468.1 [2320.5 to 78167.7]
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 26 (Day 182) post Dose 2: number analyzed (Participants) | 6
  Response antibody titers IgG S Protein reference strain (ELISA) - Week 26 (Day 182) post Dose 2 | 10833.5 [1763.7 to 66543.9]

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events: within 7 days after each IMP dose; SAEs: from Day 1 (Dose 1) up to Day 182 after Dose 2 (approximately 26 weeks after Dose 2); Other AEs in participants with Dose 2 (Group B): All AEs from Day 1 up to Day 50 and in addition if assessed as IMP-related from Day 50 up to Day 182 after Dose 2; Other AEs in participants without Dose 2 (Group A): All AEs from Day 1 up to Day 29 and in addition if assessed as IMP-related from Day 29 up to Day 182.
Description: Participants of the Group B immunology subset are also included in the respective Group B arms and therefore counted in more than one arm/group. The 'Total' arms include all participants from the respective Group A, Group B, and Group B immunology subset arms presented. Overall a total of 137 participants were enrolled into this study (including the Group B immunology subset participants).
Arm/Group | Group A Comirnaty | Group A BNT162b2s01 | Group A Total | Group B Non-transplant Participants | Group B Transplant Participants | Group B Total | Group B Immunology Subset Non-transplant Participants | Group B Immunology Subset Transplant Participants | Group B Immunology Subset Total
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/44 | 0/65 | 0/61 | 0/11 | 0/72 | 0/22 | 0/11 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/44 | 2/65 | 1/61 | 4/11 | 5/72 | 0/22 | 4/11 | 4/33
Other Adverse Events (participants affected / at risk) | 3/21 | 7/44 | 10/65 | 4/61 | 7/11 | 11/72 | 4/22 | 7/11 | 11/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A Comirnaty (N=21) | Group A BNT162b2s01 (N=44) | Group A Total (N=65) | Group B Non-transplant Participants (N=61) | Group B Transplant Participants (N=11) | Group B Total (N=72) | Group B Immunology Subset Non-transplant Participants (N=22) | Group B Immunology Subset Transplant Participants (N=11) | Group B Immunology Subset Total (N=33)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Shunt blood flow excessive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A Comirnaty (N=21) | Group A BNT162b2s01 (N=44) | Group A Total (N=65) | Group B Non-transplant Participants (N=61) | Group B Transplant Participants (N=11) | Group B Total (N=72) | Group B Immunology Subset Non-transplant Participants (N=22) | Group B Immunology Subset Transplant Participants (N=11) | Group B Immunology Subset Total (N=33)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4 | 1 | 3 | 4 | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04949490/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT04949490/SAP_001.pdf